CLINICAL TRIAL: NCT03827408
Title: Nebulized Midazolam, Dexmedetomidine, and Their Combination in Sedation of Preschoolers Undergoing Dental Treatment: A Randomized Clinical Trial
Brief Title: Nebulized Midazolam, Dexmedetomidine, and Their Combination in Sedation of Preschoolers Undergoing Dental Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Clinical Instructor, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IORG0008839
Record Dates: First submitted 2019-01-22; First posted 2019-02-01 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Dental Anxiety
Keywords: Nebulized Dexmedetomidine; Nebulized Midazolam; Moderate sedation; Dental procedural sedation; Pediatric dentistry
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated into 3 groups that will undergo a procedural sedation session via a nebulizer. Children of group I will receive nebulized solution of 0.5 mg/kg Midazolam, Group II will receive nebulized solution of 5µg/kg Dexmedetomidine, and Group III will receive a nebulized solution of 0.3 mg/kg Midazolam and 3µg/kg Dexmedetomidine respectively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The researcher, statistician and participants will be blinded to the intervention group. Only the supervisor and the anesthesiologist will be aware of the allocation group. After data collection is completed, the randomization code will be broken to reveal the allocation group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Midazolam group (MDZ) (Active Comparator): Twenty four pediatric dental patients will receive a procedural sedation session, using Nebulized solution of 0.5 mg/kg Midazolam.
  Interventions: Drug: Midazolam group (MDZ)
- Dexmedetomidine group (DEX) (Experimental): Twenty four pediatric dental patients will receive a procedural sedation session, using Nebulized solution of 5µg/kg Dexmedetomidine.
  Interventions: Drug: Dexmedetomidine group (DEX)
- Combination of Midazolam and Dexmedetomidine (MDZ/DEX) (Experimental): Twenty four pediatric dental patients will receive a procedural sedation session, using Nebulized solution of 0.3 mg/kg Midazolam, and 3µg/kg Dexmedetomidine respectively.
  Interventions: Drug: Combination of Midazolam and Dexmedetomidine (MDZ/DEX)

INTERVENTIONS:
Drug: Midazolam group (MDZ) — IV Ampules of Dormicum 15mg/ 3ml, Hoffman-La Rouche Ltd., Basel, Switzerland
  Arms: Midazolam group (MDZ)
Drug: Dexmedetomidine group (DEX) — IV Ampules of Precedex 4mcg/ml, Hospira. Inc., Lake Forest,IL USA.
  Arms: Dexmedetomidine group (DEX)
Drug: Combination of Midazolam and Dexmedetomidine (MDZ/DEX) — Combination of Nebulized solution of 0.3 mg/kg Midazolam, and 3µg/kg Dexmedetomidine respectively.(
  Arms: Combination of Midazolam and Dexmedetomidine (MDZ/DEX)

SUMMARY:
The aim of the study is to evaluate the effect of nebulized Midazolam, Dexmedetomidine, and their combination as procedural, moderate sedative agents in preschoolers undergoing dental treatment.

DETAILED DESCRIPTION:
Dental anxiety and fear related behaviors are global problems in Pediatric Dentistry. Preschoolers represent a dental behavior management problem and there is always a debate over the best behavioral management technique for preschoolers undergoing dental treatment. Moderate sedation is considered as an acceptable option.

Children who need treatment under local anesthesia, for thirty minutes will be included in the study. A total of 72 uncooperative pediatric dental patients, of age range 4-6 years, will be selected from the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University, Egypt. The participants will be randomly allocated into 3 groups that will undergo a procedural sedation session via a nebulizer. Children of group I will receive nebulized solution of 0.5 mg/kg Midazolam, Group II will receive nebulized solution of 5µg/kg Dexmedetomidine, and Group III will receive a nebulized solution of 0.3 mg/kg Midazolam and 3µg/kg Dexmedetomidine respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age range 4-6 years
* Frankl scale score 2.
* ASA I or II physical status.
* Dental intervention under local anesthesia not requiring more than 30 minutes.
* No previous dental experience.
* Parent/guardian"s written consent.

Exclusion Criteria:

* Dental treatment indicated under general anesthesia.
* Presence of facial deformities.
* History of neurological or cognitive alterations.
* Mouth breathers.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
Facemask acceptance during drug delivery | during the sedation procedure
  It will be evaluated according to Zanaty & Metainy as: poor (terrified, crying and combative), fair (moderate fear of mask not calmed with reassurance), good (slight fear of mask, easily reassured) or excellent (unafraid, cooperative and accepts mask readily)
Effect of sedation on children's future behavior | after one week in the follow-up session
  Each child's behavior will be reassessed in the follow-up sessions and compared to that at baseline (before dental treatment) using Frankl scale (ranges from 0-4)
The 'ease of treatment completion' sing separate five-point scales. | immediately after completion of the dental treatment procedures.
  This will be measured using separate five-point scales according to Surendar et al: Score 5 indicates an excellent quiet and cooperative child while score 1 indicates Prohibitive active resistance and crying; treatment cannot be rendered.
Post-operative effects of the sedation | immediately after completion of the dental treatment procedures.
  This will be assessed according to Modified Vernon et al.
Analgo-sedative effect of each drug | during the sedation procedure (time taken from drug administration till reaching satisfactory sedation)
  Onset of Sedation from drug administration until the onset of satisfactory sedation
Analgo-sedative effect of each drug | during the sedation procedure (after drug administration until reaching satisfactory sedation)
  Sedation level using Modified Observer's Assessment of Alertness/Sedation Scale. The scale is composed of 4 categories (each has scores ranging from 1-5). The categories are responsiveness, speech, facial expression and eyes. The final score is the sum of scores: the totally awake score is 20/20 and the deeply sedated score is 9/20
Analgo-sedative effect of each drug | during local anesthesia injection to start the operative procedure
  The analgesic effect of the sedative drugs will be assessed using "Face, Legs, Activity, Cry, Consolability" scale (FLACC). The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.
Analgo-sedative effect of each drug | during the sedation procedure (from its onset till meeting discharge criteria)
  The duration of sedation: defined as the onset of satisfactory sedation until the time of meeting discharge criteria according to the American Academy of Pediatric Dentistry.
Analgo-sedative effect of each drug. | during the sedation procedure (from its onset till meeting discharge criteria)
  Assessment of the most common procedural side effects such as (hypoxia, respiratory depression, agitation, arrhythmia, bradycardia, hypotension or hypertension, shivering, nausea and vomiting) will be recorded.
Amnesic effect of sedative agents. | immediately after completion of the dental treatment procedures.
  Anterograde amnesia: will be assessed according to a modification of Bulach et al.
Hemodynamic response of sedative agents. | during the sedation procedure (from its onset till meeting discharge criteria)
  Vital sign: Blood pressure (in mmHg) will be monitored using a sphygmomanometer.
Hemodynamic response of sedative agents. | during the sedation procedure (from its onset till meeting discharge criteria)
  Vital sign: Heart rate will be counted
Hemodynamic response of sedative agents. | during the sedation procedure (from its onset till meeting discharge criteria)
  Vital sign: Oxygen saturation will be monitored using an oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Amira A El-Khatib, MSc, Principal Investigator — Alexandria University; Nadia A Wahba, PhD, Study Director — Alexandria University; Karin ML Dowidar, PhD, Study Director — Alexandria University; Tamer AM Ghoneim, PhD, Study Director — Faculty of Medicine, Alexandria Univerity
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Zanaty OM, El Metainy SA. A comparative evaluation of nebulized dexmedetomidine, nebulized ketamine, and their combination as premedication for outpatient pediatric dental surgery. Anesth Analg. 2015 Jul;121(1):167-171. doi: 10.1213/ANE.0000000000000728. PMID 25822924
- [Background] Gomes HS, Miranda AR, Viana KA, Batista AC, Costa PS, Daher A, Machado GC, Sado-Filho J, Vieira LA, Correa-Faria P, Hosey MT, Costa LR. Intranasal sedation using ketamine and midazolam for pediatric dental treatment (NASO): study protocol for a randomized controlled trial. Trials. 2017 Apr 11;18(1):172. doi: 10.1186/s13063-017-1919-2. PMID 28399933
- [Background] Guideline for Monitoring and Management of Pediatric Patients Before, During, and After Sedation for Diagnostic and Therapeutic Procedures: Update 2016. Pediatr Dent. 2016 Oct 15;38(5):77-106. PMID 28206886
- [Background] Tobias JD, Leder M. Procedural sedation: A review of sedative agents, monitoring, and management of complications. Saudi J Anaesth. 2011 Oct;5(4):395-410. doi: 10.4103/1658-354X.87270. PMID 22144928
- [Background] Surendar MN, Pandey RK, Saksena AK, Kumar R, Chandra G. A comparative evaluation of intranasal dexmedetomidine, midazolam and ketamine for their sedative and analgesic properties: a triple blind randomized study. J Clin Pediatr Dent. 2014 Spring;38(3):255-61. doi: 10.17796/jcpd.38.3.l828585807482966. PMID 25095322
- [Background] Singh C, Pandey RK, Saksena AK, Chandra G. A comparative evaluation of analgo-sedative effects of oral dexmedetomidine and ketamine: a triple-blind, randomized study. Paediatr Anaesth. 2014 Dec;24(12):1252-9. doi: 10.1111/pan.12493. Epub 2014 Jul 25. PMID 25065424
- [Background] Li BL, Zhang N, Huang JX, Qiu QQ, Tian H, Ni J, Song XR, Yuen VM, Irwin MG. A comparison of intranasal dexmedetomidine for sedation in children administered either by atomiser or by drops. Anaesthesia. 2016 May;71(5):522-8. doi: 10.1111/anae.13407. Epub 2016 Mar 3. PMID 26936022
- [Background] Harbuz DK, O'Halloran M. Techniques to administer oral, inhalational, and IV sedation in dentistry. Australas Med J. 2016 Feb 29;9(2):25-32. doi: 10.4066/AMJ.2015.2543. eCollection 2016. PMID 26989448
- [Background] Greaves A. The use of Midazolam as an Intranasal Sedative in Dentistry. SAAD Dig. 2016 Jan;32:46-9. PMID 27145560
- [Background] Bulach R, Myles PS, Russnak M. Double-blind randomized controlled trial to determine extent of amnesia with midazolam given immediately before general anaesthesia. Br J Anaesth. 2005 Mar;94(3):300-5. doi: 10.1093/bja/aei040. Epub 2004 Nov 26. PMID 15567810
- [Background] Silva FC, Thuler LC. Cross-cultural adaptation and translation of two pain assessment tools in children and adolescents. J Pediatr (Rio J). 2008 Jul-Aug;84(4):344-9. doi: 10.2223/JPED.1809. PMID 18688551
- [Background] Vernon DT, Schulman JL, Foley JM. Changes in children's behavior after hospitalization. Some dimensions of response and their correlates. Am J Dis Child. 1966 Jun;111(6):581-93. doi: 10.1001/archpedi.1966.02090090053003. No abstract available. PMID 5939538
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Background] Yuen VM, Hui TW, Irwin MG, Yao TJ, Chan L, Wong GL, Shahnaz Hasan M, Shariffuddin II. A randomised comparison of two intranasal dexmedetomidine doses for premedication in children. Anaesthesia. 2012 Nov;67(11):1210-6. doi: 10.1111/j.1365-2044.2012.07309.x. Epub 2012 Sep 5. PMID 22950484
- [Background] Canpolat DG, Yildirim MD, Aksu R, Kutuk N, Alkan A, Cantekin K. Intravenous ketamine, propofol and propofol-ketamine combination used for pediatric dental sedation: A randomized clinical study. Pak J Med Sci. 2016 May-Jun;32(3):682-7. doi: 10.12669/pjms.323.9834. PMID 27375714
- See also: American Society of Anesthesiologists. ASA Physical Status Classification System. — http://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system